CLINICAL TRIAL: NCT00077311
Title: A Phase II Randomized Study Of Dose-Dense Docetaxel And Cisplatin Every Two Weeks With Pegfilgrastim And Darbepoetin Alfa With And Without The Chemoprotector BNP7787 In Patients With Advanced Non-Small Cell Lung Cancer
Brief Title: Docetaxel and Cisplatin With or Without Dimesna in Treating Patients With Stage IIIB or Stage IV Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CALGB-30303; U10CA031946 (NIH); CALGB-30303; CDR0000350089 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2004-02-10; First posted 2004-02-12 (Estimated); Last update posted 2016-06-30 (Estimated); Status verified 2016-06

CONDITIONS: Anemia; Drug/Agent Toxicity by Tissue/Organ; Lung Cancer; Neutropenia
Keywords: drug/agent toxicity by tissue/organ; anemia; neutropenia; stage IV non-small cell lung cancer; stage IIIB non-small cell lung cancer; recurrent non-small cell lung cancer; squamous cell lung cancer; large cell lung cancer; adenocarcinoma of the lung; bronchoalveolar cell lung cancer; adenosquamous cell lung cancer
MeSH Terms: conditions — Anemia; Drug-Related Side Effects and Adverse Reactions; Lung Neoplasms; Neutropenia; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma of Lung; Adenocarcinoma, Bronchiolo-Alveolar | interventions — Darbepoetin alfa; pegfilgrastim; Cisplatin; Docetaxel; 2,2'-dithiodiethanesulfonic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Chemotherapy without BNP7787 (Experimental): Chemotherapy with dose-dense docetaxel and cisplatin with pegfilgrastim and darbepoetin for pts with NSCLC
  Interventions: Biological: darbepoetin alfa; Biological: pegfilgrastim; Drug: cisplatin; Drug: docetaxel
- Chemotherapy + BNP7787 (Experimental): Chemotherapy with dose-dense docetaxel and cisplastin with pegfilgrastim and darbepoetin with the addition of BNP7787
  Interventions: Biological: darbepoetin alfa; Biological: pegfilgrastim; Drug: cisplatin; Drug: docetaxel; Drug: BNP7787

INTERVENTIONS:
Biological: darbepoetin alfa — 200 mcg sub Q on day 1 of each cycle if HgB < or = 11 g/dL
Biological: pegfilgrastim — 6 mg sub Q day 2 of each cycle
Drug: cisplatin — 75 mg/sq m IV over 1 hr Day 1 of each cycle
Drug: docetaxel — 75 mg/sq m IV over 1 hr Day 1 of each cycle
Drug: BNP7787 — 40 g IV over 30 min Day 1 of each cycle
  Arms: Chemotherapy + BNP7787

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as docetaxel and cisplatin, work in different ways to stop tumor cells from dividing so they stop growing or die. Chemoprotective drugs, such as dimesna, may help prevent or decrease the side effects (such as nerve, kidney, and inner ear damage) caused by chemotherapy.

PURPOSE: This randomized phase II trial is studying giving docetaxel and cisplatin together with dimesna to see how well it works compared to giving docetaxel and cisplatin alone in treating patients with stage IIIB or stage IV non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the incidence and severity of peripheral neuropathy in patients with stage IIIB or IV non-small cell lung cancer treated with docetaxel and cisplatin with or without dimesna.
* Compare the feasibility of these regimens, in terms of febrile neutropenia and treatment delays, in these patients.
* Compare the objective response rate in patients treated with these regimens.

Secondary

* Compare the survival and failure-free survival of patients treated with these regimens.
* Compare the toxicity profile of these regimens in these patients.
* Compare the incidence and severity of cisplatin-induced nephrotoxicity in patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are randomized to 1 of 2 treatment arms.

* Arm I*: Patients receive docetaxel IV over 1 hour and cisplatin IV over 1 hour on day 1 and pegfilgrastim subcutaneously (SC) on day 2.
* Arm II*: Patients receive docetaxel, cisplatin, and pegfilgrastim as in arm I and dimesna IV over 30 minutes on day 1.

NOTE: *In both arms, darbepoetin alfa is administered SC on day 1 of each course for hemoglobin ≤ 11 g/dL.

In both arms, treatment repeats every 2 weeks for a total of 6 courses in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 1 year and then every 6 months for 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed* non-small cell lung cancer of 1 of the following subtypes:

  * Squamous carcinoma
  * Basaloid carcinoma
  * Adenocarcinoma
  * Bronchoalveolar carcinoma
  * Adenosquamous carcinoma
  * Large cell carcinoma
  * Large cell neuroendocrine carcinoma
  * Giant cell carcinoma
  * Sarcomatoid carcinoma
  * Non-small cell carcinoma not otherwise specified NOTE: *Histologic or cytologic confirmation of recurrence is required for patients who have undergone prior complete resection
* Stage IIIB disease due to malignant pleural effusion OR stage IV disease
* Measurable disease

  * At least 1 unidimensionally measurable lesion at least 20 mm by conventional techniques OR at least 10 mm by spiral CT scan
  * The following are considered nonmeasurable disease:

    * Bone lesions
    * Brain metastases or leptomeningeal disease
    * Ascites
    * Pleural/pericardial effusion
    * Abdominal masses not confirmed and followed by imaging techniques
    * Cystic lesions
    * Tumor lesions situated in a previously irradiated area
* Brain metastases are allowed provided patient is neurologically stable and off steroids

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-1

Life expectancy

* Not specified

Hematopoietic

* Granulocyte count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3

Hepatic

* Bilirubin ≤ 1.5 mg/dL
* AST ≤ 1.5 times upper limit of normal (ULN)
* Alkaline phosphatase ≤ 2.5 times ULN

Renal

* Creatinine ≤ ULN

Other

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No grade 2 or greater neuropathy

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No other concurrent growth factors

Chemotherapy

* No prior chemotherapy
* No other concurrent chemotherapy

Endocrine therapy

* See Disease Characteristics
* No concurrent hormonal therapy except steroids administered for adrenal failure, hormones for non-cancer-related conditions (e.g., insulin for diabetes), or intermittent dexamethasone as an antiemetic

Radiotherapy

* See Disease Characteristics
* Prior radiotherapy allowed for brain metastases only
* No concurrent palliative radiotherapy

Surgery

* See Disease Characteristics

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2004-08; Primary Completion 2006-07 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Toxicity | 12 weeks
  Toxicity profile w/ emphasis on incidence and severity of peripheral neuropathy, febrile neutropenia, and nephrotoxicity

SECONDARY OUTCOMES:
Response | during tx,q 3 mon for 1 yr, then q 6 mon for 2 yrs
Survival | q 6 mon for 2 yrs after registration, then annually

CONTACTS AND LOCATIONS:
Overall Officials: Antonius Miller, MD, Study Chair — Wake Forest University Health Sciences
Locations (64):
- United States (64):
  - El Camino Hospital, Mountain View, California
  - Beebe Medical Center, Lewes, Delaware
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - St. Francis Hospital, Wilmington, Delaware
  - St. Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital, Canton, Illinois
  - Memorial Hospital, Carthage, Illinois
  - University of Illinois Cancer Center, Chicago, Illinois
  - Veterans Affairs Medical Center - Chicago Westside Hospital, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Louis A. Weiss Memorial Hospital, Chicago, Illinois
  - Eureka Community Hospital, Eureka, Illinois
  - Galesburg Clinic, Galesburg, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hopedale Medical Complex, Hopedale, Illinois
  - Kewanee Hospital, Kewanee, Illinois
  - McDonough District Hospital, Macomb, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Oncology Hematology Associates of Central Illinois - Ottawa, Ottawa, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology/Hematology Associates of Central Illinois, P.C., Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - St. Margaret's Hospital, Spring Valley, Illinois
  - Hematology Oncology Associates of the Quad Cities, Bettendorf, Iowa
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland
  - Veterans Affairs Medical Center - Baltimore, Baltimore, Maryland
  - Union Hospital Cancer Center at Union Hospital, Elkton MD, Maryland
  - Missouri Baptist Cancer Center, St Louis, Missouri
  - Arch Medical Services, Incorporated at Center for Cancer Care Research, St Louis, Missouri
  - Cancer Resource Center - Lincoln, Lincoln, Nebraska
  - Methodist Cancer Center at Methodist Hospital - Omaha, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - CCOP - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - New Hampshire Oncology-Hematology, PA - Hooksett, Hooksett, New Hampshire
  - Lakes Region General Hospital, Laconia, New Hampshire
  - Elliot Regional Cancer Center, Manchester, New Hampshire
  - Cancer Institute of New Jersey at the Cooper University Hospital - Voorhees, Voorhees Township, New Jersey
  - Charles R. Wood Cancer Center at Glens Falls Hospital, Glens Falls, New York
  - CCOP - Hematology-Oncology Associates of Central New York, Syracuse, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Community General Hospital of Greater Syracuse, Syracuse, New York
  - Faxton Regional Cancer Center, Utica, New York
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Lenoir Memorial Cancer Center, Kinston, North Carolina
  - Zimmer Cancer Center at New Hanover Regional Medical Center, Wilmington, North Carolina
  - Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University, Columbus, Ohio
  - Cancer Care Associates - Mercy Campus, Oklahoma City, Oklahoma
  - McLeod Regional Medical Center, Florence, South Carolina
  - Veterans Affairs Medical Center - Dallas, Dallas, Texas
  - Parkland Memorial Hospital, Dallas, Texas
  - Zale Lipshy University Hospital, Dallas, Texas
  - Simmons Comprehensive Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas
  - St. Mary's Regional Cancer Center at St. Mary's Medical Center, Huntington, West Virginia

REFERENCES:
- [Result] Miller AA, Wang XF, Gu L, Hoffman P, Khatri J, Dunphy F, Edelman MJ, Bolger M, Vokes EE, Green MR; Cancer and Leukemia Group B (CALGB). Phase II randomized study of dose-dense docetaxel and cisplatin every 2 weeks with pegfilgrastim and darbepoetin alfa with and without the chemoprotector BNP7787 in patients with advanced non-small cell lung cancer (CALGB 30303). J Thorac Oncol. 2008 Oct;3(10):1159-65. doi: 10.1097/JTO.0b013e318186fb0d. PMID 18827613